CLINICAL TRIAL: NCT03306121
Title: Phase Ⅲ Trial of Induction Chemotherapy（TPF） Followed by Concurrent Chemoradiotherapy Versus Concurrent Chemoradiotherapy Followed by Adjuvant Chemotherapy (PF) in Patients With High Risk Nasopharyngeal Carcinoma
Brief Title: TPF+CCRT vs.CCRT+PF in High Risk Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-034
Record Dates: First submitted 2017-10-01; First posted 2017-10-10 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma;Induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPF+CCRT (Experimental): Patients receive induction chemotherapy with paclitaxel liposome (135mg/m2 on day 1) ,cisplatin (25mg/m2 on day 1-3) and 5-fluorouracil (750mg/m2 civ 120h) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg/m2) concurrent every three weeks during radiotherapy (D1,D22,D43 of RT) .
  Interventions: Drug: TPF+CCRT
- CCRT+ PF (Active Comparator): Patients receive concurrent IMRT and cisplatin (100mg/m2) concurrent every three weeks during radiotherapy (D1,D22,D43 of RT) , then followed by three cycles of adjuvant chemotherapy with cisplatin (80mg/m2 on day 1) and 5-fluorouracil (1000mg/m2 civ 96h) every four weeks for three cycles four weeks after radiotherapy.
  Interventions: Drug: CCRT+ PF

INTERVENTIONS:
Drug: TPF+CCRT — Patients receive paclitaxel liposome (135mg/m2 on day 1) , cisplatin (25mg/m2 on day 1-3) and 5-fluorouracil (750mg/m2 civ 120h) every three weeks for three cycles of induction chemotherapy before radiotherapy.
  Patients receive IMRT and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy (D1,D22,D43 of RT)
  Other Names: TPF induction chemotherapy
  Arms: TPF+CCRT
Drug: CCRT+ PF — Patients receive cisplatin (80mg/m2 on day 1) and 5-fluorouracil (1000mg/m2 civ 96h) every four weeks for three cycles 4 weeks after radiotherapy.
  Patients receive IMRT and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy (D1,D22,D43 of RT)
  Other Names: Adjuvant PF
  Arms: CCRT+ PF

SUMMARY:
To see the effect of induction chemotherapy（TPF） followed by concurrent chemoradiotherapy versus concurrent chemoradiotherapy followed by adjuvant chemotherapy (PF) in treating patients with high risk nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage AnyTN2-3M0 and plasma EBV DNA≥1500copies/ml are randomly assigned to receive TPF(paclitaxel liposome+cisplatin+5-fluorouracil) induction chemotherapy plus concurrent chemoradiotherapy (investigational arm) or concurrent chemoradiotherapy plus PF (cisplatin+5-fluorouracil) adjuvant chemotherapy (control arm). Patients in both arms receive intensity-modulated radiotherapy(IMRT), and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy. Patients in the investigational arm receive paclitaxel liposome (135mg/m2 on day 1), cisplatin (25mg/m2 on day 1-3) and 5-fluorouracil (750mg/m2 civ 120h) every three weeks for three cycles before the radiotherapy. Patients in the control arm receive adjuvant cisplatin (80mg/m2 on day 1) and 5-fluorouracil (1000mg/m2 civ 96h) every four weeks for three cycles after the radiotherapy. The primary end point is progress-free survival (PFS). Secondary end points include overall survival(OS),locoregional failure-free survival(LRRFS), distant metastasis-free survival(DMFS), overall response rates after treatments and toxic effects(short-term and long-term). All efficacy analyses are conducted in the intention-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing carcinoma (according to World Health Organization (WHO) histologically type).
* Original clinical staged as anyT N2-3M0（according to the American Joint Committee on Cancer(AJCC) 7th edition）and plasma EBVDNA≥1500copies/ml
* No evidence of distant metastasis (M0).
* Age 18-65 years old.
* ECOG Performance status less or equal to 1
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age <18 or >65years.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation.
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival(LRRFS) | 3 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall response rate | 16 weeks after completion of IMRT
  Tumour response was classified according to RECIST, version 1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria.Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang Mai, MD,PhD, Study Chair — Sun Yat-sen Universitty Cancer Center
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Result] Lee AW, Tung SY, Ngan RK, Chappell R, Chua DT, Lu TX, Siu L, Tan T, Chan LK, Ng WT, Leung TW, Fu YT, Au GK, Zhao C, O'Sullivan B, Tan EH, Lau WH. Factors contributing to the efficacy of concurrent-adjuvant chemotherapy for locoregionally advanced nasopharyngeal carcinoma: combined analyses of NPC-9901 and NPC-9902 Trials. Eur J Cancer. 2011 Mar;47(5):656-66. doi: 10.1016/j.ejca.2010.10.026. Epub 2010 Nov 26. PMID 21112774
- [Result] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Result] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Result] Chen C, Wang FH, An X, Luo HY, Wang ZQ, Liang Y, Zhang L, Li YH. Triplet combination with paclitaxel, cisplatin and 5-FU is effective in metastatic and/or recurrent nasopharyngeal carcinoma. Cancer Chemother Pharmacol. 2013 Feb;71(2):371-8. doi: 10.1007/s00280-012-2020-x. Epub 2012 Nov 10. PMID 23143190
- [Derived] Guo SS, Li XY, Liu LT, Jia GD, Liu SL, Sun XS, Luo DH, Yang JH, Xie SY, Li YF, Lv X, Xiang YQ, Xia WX, Sun R, Liu Q, Li JB, Wang P, Yang Q, Wang L, Wen DX, Jin J, Lin JY, Mo HY, Guo L, Zhao C, Guo X, Chen QY, Tang LQ, Mai HQ. Induction vs Adjuvant Chemoradiotherapy in Patients With High-Risk N2 to N3 Nasopharyngeal Carcinoma: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2025 Aug 1;11(8):864-873. doi: 10.1001/jamaoncol.2025.1597. PMID 40531520